CLINICAL TRIAL: NCT00658957
Title: A Phase II, Randomized, Parallel, Double-blind, Placebo-controlled Study to Assess Prevention of Infection Using a Topical Gentamicin-Collagen Sponge in Diabetic Patients With Uninfected Lower Extremity Skin Ulcers
Brief Title: Prevention of Infection Using a Topical Gentamicin-Collagen Sponge in Diabetic Patients With An Uninfected Foot Ulcer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Innocoll (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: INN-TOP-002
Record Dates: First submitted 2008-04-10; First posted 2008-04-16 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetes; Foot Ulcer
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Foot Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Daily standard wound care and topical application of the gentamicin-collagen sponge twice weekly
  Interventions: Drug: gentamicin-collagen sponge
- B (Placebo Comparator): Daily standard wound care and topical application of the placebo sponge twice weekly
  Interventions: Drug: placebo collagen sponge

INTERVENTIONS:
Drug: gentamicin-collagen sponge — 5 × 5 cm sponge
  Other Names: Collatamp G
  Arms: A
Drug: placebo collagen sponge — 5 × 5 cm sponge
  Arms: B

SUMMARY:
The purpose of this study is to determine the safety and efficacy of the topical gentamicin collagen sponge (gentamicin sponge) combined with standard of care (daily wound care, off-loading, diabetic control and debridement by a physician or podiatrist), compared with placebo sponge combined with standard of care, in preventing infection of diabetic lower extremity skin ulcers.

DETAILED DESCRIPTION:
Infected skin ulcers with diabetes can be very debilitating because they are difficult to heal. Diabetic ulcers are responsible for frequent health care visits, and are a major predictor of amputation. Diabetic ulcers can be caused by a patient's inability to sense pain or warmth as well as peripheral vascular disease, which causes diminished blood flow to the foot. Early aggressive treatment is necessary to prevent infection and ultimately prevent the need for amputation.

Gentamicin is an antibiotic that is effective in treating certain kinds of infection. Collagen is a protein that is found in all mammals. The gentamicin-collagen sponge is a thin flat sponge made out of collagen that comes from cow tendons and containing gentamicin. When applied to an open ulcer, the collagen breaks down and the gentamicin is released into the ulcer, but very little is absorbed into the blood stream. The high levels of gentamicin in the open infected ulcer may help treat the infection.

In this study, all subjects will be given the necessary supplies and taught how to take care their foot ulcer. Subjects will be randomly assigned to receive either the gentamicin-collagen sponge or a plain collagen sponge. The sponge will be applied into the ulcer twice a week during the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Is a man or woman aged ≥ 18 and ≤ 80 years.
* Has diabetes mellitus according to the American Diabetes Association criteria.
* Has a single skin ulcer below the knee, defined as "uninfected" by the Infectious Disease Society of America Guidelines (Wound lacking purulence or any manifestations of inflammation).
* Has had an x-ray of the affected area within the 2 days immediately preceding or at Visit 1 (Baseline/Randomization) that is negative for osteomyelitis.
* Has an ankle-brachial index (ABI) ≥ 0.7 and ≤ 1.3. (Note: Patients with ABI < 0.7 or > 1.3 may be included if they have either a transcutaneous oxygen pressure or a toe pressure ≥ 40 mm Hg on the limb with the target ulcer.)
* Meets certain minimal laboratory criteria.
* If female, is nonpregnant (negative pregnancy tests at the Baseline/Randomization Visit) and nonlactating.
* If female, is either not of childbearing potential (defined as postmenopausal for at least 1 year or surgically sterile [bilateral tubal ligation, bilateral oophorectomy, or hysterectomy]) or practicing 1 of the following medically-acceptable methods of birth control and agrees to continue with the regimen throughout the study:

Oral, implantable or injectable contraceptives for 3 consecutive months before the Baseline/Randomization Visit.

Total abstinence from sexual intercourse (minimum of 1 complete menstrual cycle before the Baseline/Randomization Visit).

Intrauterine device (IUD). Double barrier method (condoms, sponge, diaphragm or vaginal ring with spermicidal jellies or cream).

* Willing to return to the study facility for the Posttreatment Evaluation Visit.
* Must be able to fluently speak and understand English and be able to provide meaningful written informed consent for the study.

Exclusion Criteria:

* Has a known history of hypersensitivity to gentamicin (or other systemic aminoglycosides) or any of the test article or reference product components.
* Has a known hypersensitivity to bovine collagen.
* Has any uncontrolled illnesses that, in the opinion of the Investigator, would interfere with interpreting the results of the study.
* Has a target ulcer with a wound size > 5 × 5 cm.
* Has gangrene or infection of the affected limb.
* Has a wound associated with prosthetic material or device.
* Received any topical or systemic antimicrobial therapy within the 2 weeks prior to study entry (Visit 1 [Day 1]).
* Has documented osteomyelitis.
* If severely immunocompromised, may be excluded at the discretion of the Investigator.
* Has a history of alcohol or substance abuse in the past 12 months.
* Is undergoing dialysis (renal or peritoneal) or has history of kidney transplant.
* Has history of myasthenia gravis or other neurological condition where gentamicin use is contraindicated as determined by the Investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2008-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
The percentage of patients who remain free of signs and symptoms of infection until the end of the study | Up to 3 months

SECONDARY OUTCOMES:
Time (days) to complete wound closure | Actual time
Time (days) to presence of ≥ 1 of the signs and symptoms of infection | Actual time
Absolute and percent decrease in total wound surface area | End of Study
Pathogen burden in patients who discontinue because of infection | Throughout study period
Treatment emergent Adverse Events | Throughout study period

CONTACTS AND LOCATIONS:
Overall Officials: David Prior, Study Director — Innocoll
Locations (1):
- Chesapeake Foot and Ankle Center, Pasadena, Maryland, United States